CLINICAL TRIAL: NCT00576758
Title: An Open-label, Multi-center, Randomized Study to Evaluate the Efficacy on Tumor Response of GA101 (RO5072759) Monotherapy Versus Rituximab Monotherapy in Patients With Relapsed CD20+ Indolent Non-Hodgkin's Lymphoma
Brief Title: GAUSS: A Study of Obinutuzumab (RO5072759) in Patients With Indolent Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO21003
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Results first posted 2014-03-31 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — obinutuzumab; Rituximab

ARMS (2):
- Obinutuzumab (Experimental): Participants received 1000 mg obinutuzumab intravenous (IV) infusion once a week on Days 1, 8, 15, and 22 in the Induction Period. 2 months following the last infusion, participants without disease progression, were eligible to receive a 1000 mg IV infusion every two months for 2 years in the Extension Period. All participants received oral acetaminophen/ paracetamol (1000 mg) and an antihistamine such as diphenhydramine (50-100 mg), 30-60 minutes prior to each infusion.
  Interventions: Drug: obinutuzumab (RO5072759)
- Rituximab (Active Comparator): Participants received 375 mg/m^2 rituximab IV infusion once a week on Days 1, 8, 15 and 22 in the Induction Period. 2 months following the last infusion, participants without disease progression were eligible to receive a 375 mg/m^2 rituximab IV infusion once every two months for 2 years in the Extension Period. All participants received oral acetaminophen/ paracetamol (1000 mg) and an antihistamine such as diphenhydramine (50-100 mg), 30-60 minutes prior to each infusion.
  Interventions: Drug: rituximab

INTERVENTIONS:
Drug: obinutuzumab (RO5072759) — 1000 mg obinutuzumab intravenous (IV) infusion once a week for 4 weeks.
  Other Names: RO5072759; GA101; GAZYVA®
  Arms: Obinutuzumab
Drug: rituximab — 375 mg/m^2 rituximab IV infusion once a week for 4 weeks.
  Arms: Rituximab

SUMMARY:
This study will investigate the efficacy of weekly intravenous obinutuzumab [GA101 (RO5072759)] monotherapy, in patients with relapsed CD20+ indolent Non-Hodgkin's Lymphoma. Patients will be randomized to receive either GA101 or rituximab, given as four weekly infusions. At the conclusion of the initial trial patients may be eligible to continue therapy up to 24 months. The anticipated time on study treatment is 3- 24 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age
* relapsed CD20+ indolent B-cell non-Hodgkin's lymphoma
* documented history of response of >/= 6 months duration from last rituximab-containing regimen
* clinical indication for treatment as determined by the investigator
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2

Exclusion Criteria:

* prior use of any investigational monoclonal antibody within 6 months of study start
* prior use of any anti-cancer vaccine
* prior use of rituximab within 8 weeks of study entry
* radioimmunotherapy within 3 months prior to study entry
* Central Nervous System (CNS) lymphoma or evidence of transformation to high-grade or diffuse large B-cell lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2008-01; Primary Completion 2011-09 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (62):
- United States (13):
  - Los Angeles, California
  - Denver, Colorado
  - Gainesville, Florida
  - Tampa, Florida
  - Augusta, Georgia
  - Cumberland, Maryland
  - Hackensack, New Jersey
  - New York, New York
  - Rochester, New York
  - Concord, North Carolina
  - Columbus, Ohio
  - Houston, Texas
  - Seattle, Washington
- Buenos Aires, Argentina
- Austria (3):
  - Innsbruck
  - Salzburg
  - Vienna
- Belgium (3):
  - Brussels
  - Ghent
  - Mont-godinne
- Brazil (4):
  - Goiânia, Goiás
  - Porto Alegre, Rio Grande do Sul
  - Piracicaba, São Paulo
  - São Paulo, São Paulo
- Canada (5):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Kingston, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Croatia (2):
  - Rijeka
  - Zagreb
- Denmark (3):
  - Aarhus
  - Copenhagen
  - Vejle
- Greece (2):
  - Athens
  - Thessaloniki
- Italy (7):
  - Bologna
  - Brescia
  - Milan
  - Novara
  - Pisa
  - Reggio Calabria
  - Rozzano
- Netherlands (3):
  - Amsterdam
  - Groningen
  - Rotterdam
- Warsaw, Poland
- Spain (8):
  - Palma de Mallorca, Balearic Islands
  - Barcelona, Barcelona
  - A Coruña, La Coruña
  - Madrid, Madrid
  - Salamanca, Salamanca
  - Seville, Sevilla
  - Valencia, Valencia
  - Zaragoza, Zaragoza
- Sweden (2):
  - Huddinge
  - Malmo
- Switzerland (2):
  - Sankt Gallen
  - Zurich
- Turkey (Türkiye) (2):
  - Istanbul
  - Izmir
- London, United Kingdom

REFERENCES:
- [Derived] Gibiansky E, Gibiansky L, Buchheit V, Frey N, Brewster M, Fingerle-Rowson G, Jamois C. Pharmacokinetics, exposure, efficacy and safety of obinutuzumab in rituximab-refractory follicular lymphoma patients in the GADOLIN phase III study. Br J Clin Pharmacol. 2019 Sep;85(9):1935-1945. doi: 10.1111/bcp.13974. Epub 2019 Jul 12. PMID 31050355
- [Derived] Kostakoglu L, Goy A, Martinelli G, Caballero D, Crump M, Gaidano G, Baetz T, Buckstein R, Fine G, Fingerle-Rowson G, Berge C, Sahin D, Press O, Sehn L. FDG-PET is prognostic and predictive for progression-free survival in relapsed follicular lymphoma: exploratory analysis of the GAUSS study. Leuk Lymphoma. 2017 Feb;58(2):372-381. doi: 10.1080/10428194.2016.1196815. Epub 2016 Jun 24. PMID 27339738
- [Derived] Sehn LH, Goy A, Offner FC, Martinelli G, Caballero MD, Gadeberg O, Baetz T, Zelenetz AD, Gaidano G, Fayad LE, Buckstein R, Friedberg JW, Crump M, Jaksic B, Zinzani PL, Padmanabhan Iyer S, Sahin D, Chai A, Fingerle-Rowson G, Press OW. Randomized Phase II Trial Comparing Obinutuzumab (GA101) With Rituximab in Patients With Relapsed CD20+ Indolent B-Cell Non-Hodgkin Lymphoma: Final Analysis of the GAUSS Study. J Clin Oncol. 2015 Oct 20;33(30):3467-74. doi: 10.1200/JCO.2014.59.2139. Epub 2015 Aug 17. PMID 26282650
- [Derived] Sehn LH, Assouline SE, Stewart DA, Mangel J, Gascoyne RD, Fine G, Frances-Lasserre S, Carlile DJ, Crump M. A phase 1 study of obinutuzumab induction followed by 2 years of maintenance in patients with relapsed CD20-positive B-cell malignancies. Blood. 2012 May 31;119(22):5118-25. doi: 10.1182/blood-2012-02-408773. Epub 2012 Mar 20. PMID 22438256

RESULTS

PARTICIPANT FLOW:
Period: Induction Treatment Period
Arm/Group | Rituximab | Obinutuzumab
Started | 87 | 88
Received Treatment | 86 | 87
Completed | 79 | 83
Not Completed | 8 | 5
Not completed — Adverse event or Intercurrent illness | 3 | 3
Not completed — Insufficient therapeutic response | 2 | 0
Not completed — Violation of selection criteria at entry | 1 | 1
Not completed — Death | 1 | 0
Not completed — Refused treatment/ Did not Cooperate | 0 | 1
Not completed — Withdrew consent | 1 | 0
Period: Extension Treatment Period
Arm/Group | Rituximab | Obinutuzumab
Started | 72 (6 patients did not enter extended treatment phase/follow-up + 1 patient entered follow-up.) | 73 (8 patients did not enter extended treatment phase/follow-up phase + 2 patients entered follow-up.)
Completed | 30 (+ 2 patients (pts) who withdrew prior to receiving study drug.) | 30
Not Completed | 42 | 43
Not completed — Adverse event or Intercurrent illness | 6 | 7
Not completed — Death | 1 | 1
Not completed — Refused treatment/did not cooperate | 2 | 1
Not completed — Insufficient therapeutic response | 30 | 33
Not completed — Administrative/Other | 3 | 1
Period: Follow-up Period
Arm/Group | Rituximab | Obinutuzumab
Started | 55 (Includes 23 pts who entered follow-up after induction and didn't enter the extended treatment phase.) | 51 (Includes 21 pts who entered follow-up after induction and didn't enter the extended treatment phase.)
Completed | 28 | 34
Not Completed | 27 | 17
Not completed — Administrative/Other | 6 | 8
Not completed — Death | 3 | 3
Not completed — Insufficient therapeutic response | 16 | 5
Not completed — Withdrew consent | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab | Obinutuzumab | Total
Number analyzed (Participants) | 87 | 88 | 175
Age, Customized [Number; unit: participants]
  <65 years | 49 | 47 | 96
  65-70 years | 22 | 22 | 44
  >70 years | 16 | 19 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 42 | 85
  Male | 44 | 46 | 90

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Response At the End of Induction Period
Description: Overall response was defined as Complete Response (CR), Complete Response/Unconfirmed (CRu) or Partial Response (PR) as assessed by investigator at end of induction treatment. Computed tomography imaging was used for the primary assessment of tumor response per 1999 criteria by Cheson.
  CR was defined as the disappearance of all clinical and radiographic evidence of disease, disease-related symptoms and normalization of biochemical abnormalities of NHL.
  CRu was CR plus one or more of the following: A residual lymph node mass greater than 1.5 cm in greatest transverse diameter that has regressed by more than 75% in the sum of the products of the greatest diameter (tumors)(SPD) and/or indeterminate bone marrow.
  PR was defined as 50% decrease in SPD of the 6 largest dominant nodes or nodal masses. No increase in the size of the other nodes, liver, or spleen. Splenic and hepatic nodules must regress by at least 50% in the SPD. No new sites of disease.
Time Frame: Randomization to clinical cutoff: 01 September 2011 (Up to 70 days)
Population: Participants from the Intent-to-treat (ITT) population (all randomized participants) with follicular non-Hodgkin's lymphoma (NHL) at the time of diagnosis.
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab | Obinutuzumab
Number analyzed (Participants) | 75 | 74
Percentage of participants | 33.3 | 44.6
Statistical Analysis 1: Comparison: Rituximab vs Obinutuzumab; Test type: Superiority or Other; p = 0.1587, Chi-squared; Mean Difference (Final Values) = 11.26, 60% CI 2-sided [3.9 to 18.7]

2. Secondary Outcome: Percentage of Participants With Complete Response at the End of the Induction Period
Description: Computed tomography imaging was used for the primary assessment of tumor response per 1999 criteria by Cheson. CR is defined as the disappearance of all clinical and radiographic evidence of disease, disease-related symptoms and normalization of biochemical abnormalities of NHL. All lymph nodes and nodal masses must have regressed to normal size. The spleen, if considered to be enlarged before therapy on the basis of a CT scan, must have regressed in size and must not be palpable on physical examination. Any macroscopic nodules in any organs detectable on imaging techniques should no longer be present. Other organs considered to be enlarged before therapy due to involvement by lymphoma, such as liver and kidneys, must have decreased in size. If the bone marrow was involved by lymphoma before treatment, the infiltrate must be cleared on repeat bone marrow aspirate and biopsy of the same site.
Time Frame: Randomization to clinical cutoff : 01 September 2011 (Up to 70 days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rituximab | Obinutuzumab
Number analyzed (Participants) | 75 | 74
Percentage of participants | 5.3 [1.5 to 13.1] | 12.2 [5.7 to 21.8]
Statistical Analysis 1: Comparison: Rituximab vs Obinutuzumab; Test type: Superiority or Other; Mean Difference (Final Values) = 6.83, 95% CI 2-sided [-2.9 to 16.6]

3. Secondary Outcome: Percentage of Participants With Partial Response (PR) at the End of the Induction Period
Description: Computed tomography imaging was used for the primary assessment of tumor response per 1999 criteria by Cheson. PR was defined as 50% decrease in SPD of the 6 largest dominant nodes or nodal masses. No increase in the size of the other nodes, liver, or spleen. Splenic and hepatic nodules must regress by at least 50% in the SPD. No new sites of disease.
Time Frame: Randomization to clinical cutoff : 01 September 2011 (Up to 70 days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rituximab | Obinutuzumab
Number analyzed (Participants) | 75 | 74
Percentage of participants | 28.0 [18.2 to 39.6] | 32.4 [22.0 to 44.3]

4. Secondary Outcome: Percentage of Participants With Best Overall Response Achieved at Any Time During the Study Treatment
Description: Overall response was defined as Complete Response (CR), Complete Response/Unconfirmed (CRu) or Partial Response (PR) as assessed by investigators during study treatment (induction or extended treatment phase). Computed tomography imaging was used for the primary assessment of tumor response per 1999 criteria by Cheson.
  CR was defined as the disappearance of all clinical and radiographic evidence of disease, disease-related symptoms and normalization of biochemical abnormalities of NHL.
  CRu was CR plus one or more of the following: A residual lymph node mass greater than 1.5 cm in greatest transverse diameter that has regressed by more than 75% in the sum of the products of the greatest diameter (tumors)(SPD) and/or indeterminate bone marrow.
  PR was defined as 50% decrease in SPD of the 6 largest dominant nodes or nodal masses. No increase in the size of the other nodes, liver, or spleen. Splenic and hepatic nodules must regress by at least 50% in the SPD. No new sites of disease.
Time Frame: Randomization to clinical cutoff : 01 September 2011 (Up to 70 days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rituximab | Obinutuzumab
Number analyzed (Participants) | 75 | 74
Percentage of participants
  Complete Response | 18.7 [10.6 to 29.3] | 35.1 [24.4 to 47.1]
  Partial Response | 45.3 [33.8 to 57.3] | 31.1 [20.8 to 42.9]
  Stable Disease | 26.7 [17.1 to 38.1] | 21.6 [12.9 to 32.7]
  Progressive Disease | 5.3 [1.5 to 13.1] | 8.1 [3.0 to 16.8]

5. Secondary Outcome: Number of Participants With Improved Overall Response During the Extended Treatment Period
Description: Overall response was defined as Complete Response (CR), Complete Response/Unconfirmed (CRu) or Partial Response (PR) as assessed by investigators at end of induction treatment. Computed tomography imaging was used for the primary assessment of tumor response per 1999 criteria by Cheson.
Time Frame: Randomization to Clinical cutoff: 07 March 2013 (Up to 43.2 months)
Population: Participants from the Intent-to-treat (ITT) population (all randomized participants) with follicular non-Hodgkin's lymphoma (NHL) at the time of diagnosis who received treatment in the extension period.
Measure: Number; unit: Participants
Arm/Group | Rituximab | Obinutuzumab
Number analyzed (Participants) | 63 | 62
Participants | 31 | 32

6. Secondary Outcome: Percentage of Participants With Best Overall Response Achieved at Any Time During the Study Treatment
Description: as for outcome 4
Time Frame: Randomization to Clinical cutoff: 07 March 2013 (Up to 43.2 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rituximab | Obinutuzumab
Number analyzed (Participants) | 75 | 74
Percentage of participants
  Complete Response | 22.7 [13.8 to 33.8] | 41.9 [30.5 to 53.9]
  Partial Response | 41.3 [30.1 to 53.3] | 24.3 [15.1 to 35.7]
  Stable Disease | 26.7 [17.1 to 38.1] | 21.6 [12.9 to 32.7]
  Progressive Disease | 5.3 [1.5 to 13.1] | 8.1 [3.0 to 16.8]
  No Response Assessment | 4.0 [NA to NA] — Not estimable. | 4.1 [NA to NA] — Not estimable.
Statistical Analysis 1: Comparison: Rituximab vs Obinutuzumab; Test type: Superiority or Other; Mean Difference (Final Values) = 2.22, 95% CI 2-sided [-13.9 to 18.3]

7. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from randomization to the first occurrence of progression, relapse, or death from any cause as assessed by the Investigator.
  Progression was defined as a ≥ 50% increase from nadir in the SPD of any previously identified abnormal node and/or the appearance of any new lesion during or at the end of therapy.
  Relapse was defined as the appearance of any new lesion or increase by ≥ 50% in the size of previously involved sites and/or a ≥ 50% increase in greatest diameter of any previously identified node greater than 1 cm in its short axis or in the SPD of more than one node.
Time Frame: Randomization to Clinical cutoff: 07 March 2013 (Up to 43.2 months)
Population: ITT population included all randomized participants with follicular non-Hodgkin's lymphoma at the time of diagnosis. If no PFS even occurred, PFS was censored at the date of the last tumor assessment. If no tumor assessment was available patient was censored at the date of the first study drug administration.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Rituximab | Obinutuzumab
Number analyzed (Participants) | 75 | 74
Days | 772 [425 to 867] | 536 [394 to NA] — Upper limit was not estimable due to insufficient number of participants with events therefore the upper confidence limit of the survival curve is above 50%.
Statistical Analysis 1: Comparison: Rituximab vs Obinutuzumab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.62 to 1.44]

8. Secondary Outcome: Percentage of Participants With Progression-Free Survival (PFS) Events
Description: The percentage of participants with progression, relapse, or death events from any cause as assessed by the Investigator.
  Progression was defined as a ≥ 50% increase from nadir in the SPD of any previously identified abnormal node and/or the appearance of any new lesion during or at the end of therapy.
  Relapse was defined as the appearance of any new lesion or increase by ≥ 50% in the size of previously involved sites and/or a ≥ 50% increase in greatest diameter of any previously identified node greater than 1 cm in its short axis or in the SPD of more than one node.
Time Frame: Randomization to Clinical cutoff: 07 March 2013 (Up to 43.2 months)
Population: Participants from the ITT population (all randomized participants) with follicular non-Hodgkin's lymphoma at the time of diagnosis. If event did not occur, PFS was censored at the date of the last tumor assessment. If no tumor assessment is available patient was censored at the date of the first study drug administration.
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab | Obinutuzumab
Number analyzed (Participants) | 75 | 74
Percentage of participants | 57.7 | 51.4

9. Secondary Outcome: Event Free Survival
Description: Event-free survival (EFS) was defined as the time between date of randomization and the date of disease progression/relapse, death, or start of a new anti-leukemic therapy.
  Progression was defined as a ≥ 50% increase from nadir in the SPD of any previously identified abnormal node and/or the appearance of any new lesion during or at the end of therapy.
  Relapse was defined as the appearance of any new lesion or increase by ≥ 50% in the size of previously involved sites and/or a ≥ 50% increase in greatest diameter of any previously identified node greater than 1 cm in its short axis or in the SPD of more than one node.
Time Frame: Randomization to Clinical cutoff: 07 March 2013 (Up to 43.2 months)
Population: ITT population included all randomized participants with follicular non-Hodgkin's lymphoma at the time of diagnosis. If no EFS event occurred, EFS was censored at the date of the last tumor assessment. If no tumor assessment is available patient was censored at the date of the first study drug administration.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Rituximab | Obinutuzumab
Number analyzed (Participants) | 75 | 74
Days | 472.0 [362 to 772] | 472.0 [318 to 605]
Statistical Analysis 1: Comparison: Rituximab vs Obinutuzumab; Test type: Superiority or Other; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.67 to 1.50]

10. Secondary Outcome: Percentage of Participants With Event Free Survival (EFS) Events
Description: Percentage of participants with Event Free Events: disease progression/relapse, death, or start of a new anti-leukemic therapy.
  Progression was defined as a ≥ 50% increase from nadir in the SPD of any previously identified abnormal node and/or the appearance of any new lesion during or at the end of therapy.
  Relapse was defined as the appearance of any new lesion or increase by ≥ 50% in the size of previously involved sites and/or a ≥ 50% increase in greatest diameter of any previously identified node greater than 1 cm in its short axis or in the SPD of more than one node.
Time Frame: Randomization to Clinical cutoff: 07 March 2013 (Up to 43.2 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab | Obinutuzumab
Number analyzed (Participants) | 75 | 74
Percentage of participants | 64.0 | 63.5

11. Secondary Outcome: Duration of Response
Description: Duration of Response was defined as the date the response, either Complete Response (CR) or Partial Response (PR), was first recorded until the date of Disease Progression or death due to any cause. Computed tomography imaging was used for the primary assessment of tumor response per 1999 criteria by Cheson.
  CR was defined as the disappearance of all clinical and radiographic evidence of disease, disease-related symptoms and normalization of biochemical abnormalities of NHL.
  PR was defined as 50% decrease in SPD of the 6 largest dominant nodes or nodal masses. No increase in the size of the other nodes, liver, or spleen. Splenic and hepatic nodules must regress by at least 50% in the SPD. No new sites of disease.
  Disease Progression was defined as a ≥ 50% increase from nadir in the SPD of any previously identified abnormal node and/or the appearance of any new lesion during or at the end of therapy.
Time Frame: Randomization to Clinical cutoff: 07 March 2013 (Up to 43.2 months)
Population: Participants from the ITT population (all randomized participants with follicular NHL at the time of diagnosis N=75/74] with response. Patients with no documented progression after CR or PR will be censored at the last tumor assessment. If no assessment available patients will be censored at the first study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Rituximab | Obinutuzumab
Number analyzed (Participants) | 48 | 49
Months | 809 [412 to NA] — Upper limit was not estimable due to insufficient number of participants with events therefore the upper confidence limit of the survival curve is above 50%. | NA [672 to NA] — Median and Upper limit was not estimable due to insufficient number of participants with events therefore the upper confidence limit of the survival curve is above 50%.

12. Secondary Outcome: Obinutuzumab Serum PK Parameter: Terminal Half-Life (t1/2)
Description: Blood was collected for Pharmacokinetic (PK) Parameters before and after dose administration of obinutuzumab in Induction Phase Cycle 4. Serum samples were sent to a central lab and were analyzed for obinutuzumab using a validated enzyme-linked immunosorbent assay (ELISA). Terminal Half-Life was calculated in days.
Time Frame: Day 22 (pre-infusion, at end of infusion, 3-6, 20-28, 66-80 hours, 6-8, 12-16, 18-24, 28-56 days post-infusion)
Population: PK Analysis Population included all participants who received obinutuzumab and had PK samples collected as per protocol. Patients with limited PK sampling time-points were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 72
days | 41.0 (28.6)

13. Secondary Outcome: Obinutuzumab Serum PK Parameter: Maximum Serum Concentration (Cmax)
Description: Blood was collected for PK Parameters before and after dose administration of obinutuzumab in Induction Phase Cycles 1, 2, 3 and 4. Serum samples were sent to a central lab and were analyzed for obinutuzumab using a validated enzyme-linked immunosorbent assay (ELISA). Cmax was calculated in micrograms/milliliter (μg/mL).
Time Frame: Day 1 (pre-infusion, at end of infusion, 3-6, 20-28, 66-80 hours post-infusion), Days 8 and 15 (pre-infusion, at end of infusion), Day 22 (pre-infusion, at end of infusion, 3-6, 20-28, 66-80 hours, 6-8, 12-16, 18-24, 28-56 days post-infusion)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 78
μg/mL
  Cycle 1 (n=74) | 292 (87.4)
  Cycle 2 (n=78) | 448 (129)
  Cycle 3 (n=77) | 561 (158)
  Cycle 4 (n=77) | 692 (213)

14. Secondary Outcome: Obinutuzumab Serum PK Parameter: Area Under the Concentration Curve (AUClast)
Description: Blood was collected for PK Parameters before and after dose administration of obinutuzumab in Induction Phase Cycle 4. Serum samples were sent to a central lab and were analyzed for obinutuzumab using a validated enzyme-linked immunosorbent assay (ELISA). AUClast was calculated in days* micrograms/milliliter (μg/mL)
Time Frame: Day 22 (pre-infusion, at end of infusion, 3-6, 20-28, 66-80 hours, 6-8, 12-16, 18-24, 28-56 days post-infusion)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 77
day*μg/mL | 23400 (10300)

15. Secondary Outcome: Obinutuzumab Serum PK Parameter: Clearance at Steady-State (CLss)
Description: Blood was collected for PK Parameters before and after dose administration of obinutuzumab in Induction Phase Cycle 4. Serum samples were sent to a central lab and were analyzed for obinutuzumab using a validated enzyme-linked immunosorbent assay (ELISA). CLsst was calculated in milliliter/day (mL/day)
Time Frame: Day 22 (pre-infusion, at end of infusion, 3-6, 20-28, 66-80 hours, 6-8, 12-16, 18-24, 28-56 days post-infusion)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mL/day
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 72
mL/day | 308 (470)

16. Secondary Outcome: Obinutuzumab Serum PK Parameter: Volume of Distribution at Steady-State (Vss)
Description: Blood was collected for PK Parameters before and after dose administration of obinutuzumab in Induction Phase Cycle 4. Serum samples were sent to a central lab and were analyzed for obinutuzumab using a validated enzyme-linked immunosorbent assay (ELISA). Vss was calculated in liters (L).
Time Frame: Day 22 (pre-infusion, at end of infusion, 3-6, 20-28, 66-80 hours, 6-8, 12-16, 18-24, 28-56 days post-infusion)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 72
Liter | 14.6 (9.8)

17. Secondary Outcome: Obinutuzumab Serum PK Parameter: Area Under the Concentration Curve Between Dosing Interval (AUCtau)
Description: Blood was collected for PK Parameters before and after dose administration of obinutuzumab in Induction Phase Cycle 4. Serum samples were sent to a central lab and were analyzed for obinutuzumab using a validated enzyme-linked immunosorbent assay (ELISA). AUCtau was calculated in days* micrograms/milliliter (μg/mL)
Time Frame: Day 22 (pre-infusion, at end of infusion, 3-6, 20-28, 66-80 hours, 6-8, 12-16, 18-24, 28-56 days post-infusion)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 77
day*μg/mL | 4370 (1340)

18. Secondary Outcome: Obinutuzumab Trough Serum Concentration (Ctrough)
Description: Blood was collected for PK Parameters before and after dose administration of obinutuzumab in Induction Phase Cycles 2, 3 and 4. Serum samples were sent to a central lab and were analyzed for obinutuzumab using a validated enzyme-linked immunosorbent assay (ELISA). Ctrough was calculated in micrograms/milliliter (μg/mL).
Time Frame: Days 8 and 15 (pre-infusion, at end of infusion), Day 22 (pre-infusion, at end of infusion, 3-6, 20-28, 66-80 hours, 6-8, 12-16, 18-24, 28-56 days post-infusion)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 78
μg/mL
  Cycle 2 (n=78) | 154 (62.7)
  Cycle 3 (n=77) | 301 (119)
  Cycle 4 (n=75) | 418 (147)

19. Secondary Outcome: Number of Participants With Peripheral Blood B-Cell Depletion
Description: Blood was collected and sent to a central laboratory for the evaluation of cluster of differentiation 19 (CD19) by flow cytometry at the end of the induction period. B-cell depletion was defined as a CD19 result 5 % of the Baseline value after at least one dose of study drug was administered.
Time Frame: Day 22
Population: Participants from the Safety Population, all randomized participants who received study drug, with data available for analysis.
Measure: Number; unit: Participants
Arm/Group | Rituximab | Obinutuzumab
Number analyzed (Participants) | 84 | 85
Participants | 80 | 82

20. Secondary Outcome: Number of Participants With Peripheral Blood B-Cell Recovery
Description: Blood was sent to a central laboratory for the evaluation of cluster of differentiation 19 (CD19) by flow cytometry. B-cell recovery was defined as the time point when the CD-19 values return to ≥ 50% of baseline levels. The number of participants with B-cell recovery from End of Induction (treatment) Phase to 6 months of Follow-up is reported in two categories: Recovery with Progressive Disease (PD) or Recovery without PD. PD required one of the following: 50 % increase in the absolute number of circulating lymphocytes, Appearance of new palpable lymph nodes, 50 % increase in the longest diameter of any previous site of lymphadenopathy, 50 % increase in the enlargement of the liver and/or spleen or Transformation to a more aggressive histology.
Time Frame: End of last dose + 6 Months Follow-Up
Population: Participants from the Safety Population, all randomized participants who received study drug, with previous B-Cell Depletion and B-Cell assessment at 6 Month Follow-up.
Measure: Number; unit: Participants
Arm/Group | Rituximab | Obinutuzumab
Number analyzed (Participants) | 69 | 73
Participants
  Recovery with PD | 0 | 2
  Recovery without PD | 1 | 0

21. Secondary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory result), symptom, or disease temporally associated with the use of an investigational medicinal product (IMP) or other protocol-imposed intervention, regardless of attribution. A SAE was any AE that was one of the following: fatal, life-threatening, required or prolonged inpatient hospitalization, resulted in persistent or significant disability/incapacity, a congenital anomaly/birth defect in a neonate/infant born to a mother exposed to the investigational product or considered a significant medical event by the investigator. Additional information about AEs can be found in the Adverse Event Section.
Time Frame: Randomization to Clinical cutoff: 07 March 2013 (Up to 43.2 months) [Includes all AEs reported 28 days after last dose and all Related SAEs regardless of time of last dose.]
Population: Safety Population included all randomized participants who received study drug.
Measure: Number; unit: Participants
Arm/Group | Rituximab | Obinutuzumab
Number analyzed (Participants) | 86 | 87
Participants
  AE | 74 | 83
  SAE | 17 | 21

22. Secondary Outcome: Number of Participants With Infusion Related Reactions
Description: Infusion Related Reactions were AEs that occurred during the infusion or within 24 hours of the infusion.
Time Frame: Randomization to Clinical cutoff: 07 March 2013 (Up to 43.2 months)
Population: Safety Population included all randomized participants who received at least once dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Rituximab | Obinutuzumab
Number analyzed (Participants) | 86 | 87
Participants | 44 | 70

23. Secondary Outcome: Number of Participants With Human Anti-Chimeric Antibodies (HACA)
Description: Blood was collected on Day 1 and was sent to a central laboratory for analysis of human anti-chimeric antibodies (anti-rituximab antibodies) using a validated enzyme-linked immunosorbent assay (ELISA). HACA samples were not collected for participants randomized to the rituximab arm.
Time Frame: Day 1
Population: Participants from the Safety Population, all randomized participants who received study drug, who had samples available for HACA analysis.
Measure: Number; unit: Participants
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 86
Participants | 1

24. Secondary Outcome: Number of Participants With Human Anti-Human Antibodies (HAHA)
Description: Blood was collected on Day 1 pre-infusion, during the safety follow-up for those patients who did not enter the Extension period and 6 months after the last infusion of the Extension Period if applicable. Blood was sent to a central laboratory and was tested for anti-obinutuzumab antibodies using a validated enzyme-linked immunosorbent assay (ELISA). HAHA samples were not collected for participants randomized to the rituximab arm.
Time Frame: Randomization to Clinical cutoff: 07 March 2013 (Up to 43.2 months)
Population: Safety Population included all randomized participants who received study drug.
Measure: Number; unit: Participants
Arm/Group | Obinutuzumab
Number analyzed (Participants) | 86
Participants | 0

ADVERSE EVENTS:
Time Frame: First dose of study drug to 28 days past last dose of study drug (Up to 27 Months)
Description: Safety population included all randomized patients who received at least one dose of study drug. Serious Adverse Events that occurred during treatment are reported.
Arm/Group | Rituximab | Obinutuzumab
Serious Adverse Events (participants affected / at risk) | 13/86 | 13/87
Other Adverse Events (participants affected / at risk) | 70/86 | 79/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=86) | Obinutuzumab (N=87)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 2
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 2
Cellulitis (Infections and infestations) | 1 | 0
Herpes zoster disseminated (Infections and infestations) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 2
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Hepatitis cholestatic (Hepatobiliary disorders) | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1
Diastolic dysfunction (Cardiac disorders) | 0 | 1
Chronic sinusitis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=86) | Obinutuzumab (N=87)
Neutropenia (Blood and lymphatic system disorders) | 6 | 3
Abdominal pain upper (Gastrointestinal disorders) | 6 | 2
Diarrhoea (Gastrointestinal disorders) | 7 | 7
Nausea (Gastrointestinal disorders) | 7 | 8
Asthenia (General disorders) | 5 | 6
Fatigue (General disorders) | 17 | 23
Oedema peripheral (General disorders) | 4 | 6
Pyrexia (General disorders) | 9 | 5
Bronchitis (Infections and infestations) | 3 | 7
Influenza (Infections and infestations) | 5 | 3
Nasopharyngitis (Infections and infestations) | 4 | 6
Sinusitis (Infections and infestations) | 4 | 6
Upper respiratory tract infection (Infections and infestations) | 9 | 9
Infusion related reactions (Injury, poisoning and procedural complications) | 43 | 62
Decreased appetite (Metabolism and nutrition disorders) | 3 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 5
Dizziness (Nervous system disorders) | 6 | 4
Headache (Nervous system disorders) | 7 | 8
Paraesthesia (Nervous system disorders) | 2 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 20
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 6
Hypertension (Vascular disorders) | 7 | 2
Insomnia (Psychiatric disorders) | 1 | 4
Vomiting (Gastrointestinal disorders) | 3 | 4
Rhinitis (Infections and infestations) | 4 | 4
Herpes zoster (Infections and infestations) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.